CLINICAL TRIAL: NCT01299064
Title: Transcultural Mindfulness Assessment: A Mixed Methods Analysis
Status: Completed | Type: Observational
Sponsor: Pacific University (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Michael Christopher, PhD, Associate Professor, Pacific University
Other Study IDs: 1R15AT005342-01A1 (NIH); 1R15AT005342-01A1 (NIH)
Record Dates: First submitted 2011-02-17; First posted 2011-02-18 (Estimated); Last update posted 2014-10-29 (Estimated); Status verified 2014-10

CONDITIONS: Mental Health Wellness 1
Keywords: mindfulness-based intervention; symptoms reduction; mental health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Buddhist Clergy and Laypersons

SUMMARY:
Preliminary evidence attests to the effectiveness of mindfulness-based interventions in reducing symptoms associated with a variety of medical and psychological conditions. However, research progress has been hampered by discrepancies in how mindfulness has been operationalized, assessed, and practiced. Existing contemporary assessments of mindfulness were developed exclusively by Western scientists and have exhibited questionable validity, particularly among diverse cultural groups. Operational definitions of mindfulness are essential for the development of valid measures, which in turn are necessary for investigating the mechanisms of change in mindfulness-based interventions. Therefore, the overall goal of this study is to create a mindfulness measure that is informed by the experience of mindfulness experts - Theravāda, Tibetan, and Zen Buddhist clergy and lay practitioners. To do so, this study will employ the preliminary phases of the sequential exploratory mixed methods for instrument design model. The first phase will involve conducting open-ended interviews with Theravāda, Tibetan, and Zen Buddhist clergy and lay practitioners to ascertain expert information on mindfulness and closely related Buddhist concepts. This qualitative process allows the experts to define the phenomena of interest (i.e., addresses issues of validity). In the second phase, the investigators will use the themes and specific phrases evoked during the qualitative interviews to develop items for a draft closed-ended self-report measure of mindfulness. Following completion of the research outlined in this proposal, the investigators will submit a subsequent proposal to thoroughly evaluate the psychometric properties of our draft mindfulness questionnaire in a variety of different cultures and contexts. This measure can be beneficial in clinical research by helping to elucidate the mechanisms of change in mindfulness-based psychotherapies in the United States and equally so in other cultures such as Thailand, where mindfulness and other Buddhist practices have already been integrated into mainstream mental health treatment. Therefore, our aim is to create a measure that can help improve the assessment and clinical use of mindfulness.

ELIGIBILITY:
Inclusion Criteria:

* Zen, Theravada, or Tibetan clergy
* Zen, Theravada, or Tibetan layperson with meditation experience

Exclusion Criteria:

* Under 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Buddhist clergy and laypersons
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-08; Primary Completion 2011-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Pacific University, Forest Grove, Oregon, United States